CLINICAL TRIAL: NCT03551444
Title: RECURRENCE RATE OF HEPATOCELLULAR CARCINOMA AFTER TREATMENT OF CHRONIC HEPATITIS C PATIENTS WITH DIRECT ACTING ANTIVIRALS: RANDOMIZED CONTROLLED PHASE 3 TRIAL (CAUTIOUS TRIAL)
Brief Title: Recurrence Rate of Hepatocellular Carcinoma After Treatment of Chronic Hepatits C Patients With Direct Acting Antivirals: Randomized Controlled Phase 3 Trial
Acronym: CAUTIOUS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma Sayed, Ph.D Candidate, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD353/2017
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Hepatocellular Carcinoma; Hepatitis C, Chronic
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Administration of DAA-based treatment (Arm 1) (Active Comparator): Arm 1 will be divided into 2 groups by randomization according to a 1:1 ratio into:
  Group A: Administration of DAA-based treatment after 3 months of complete remission of HCC.
  Group B: Administration of DAA-based treatment after 6 months of complete remission of HCC.
  Interventions: Drug: Administration of DAA-based treatment
- Control arm (Arm 2) (Experimental): Not receiving DAAs after complete remission of HCC and to be kept on follow-up
  Interventions: Drug: Administration of DAA-based treatment

INTERVENTIONS:
Drug: Administration of DAA-based treatment — * Antiviral therapy and treatment duration (12/24 weeks) will be indicated in each patient according to the viral genotype/subtype and the severity of liver disease, in accordance with the EASL Recommendations on Treatment of Hepatitis C 2016.
  * HCV-RNA quantification will be assessed by real-time PCR, with a limit of detection (LOD) of15 IU/mL.
  * During antiviral treatment, follow-up of the Patients will be monthly by clinical and laboratory evaluation.
  * Virological response to DAA-based treatment will be assessed by quantitative HCV-RNA at the end of treatment (EOT) and at 4 and 12 weeks after the EOT, to confirm sustained virological response (SVR).
  * SVR12 is defined as undetectable HCV-RNA at week 12 after the EOT.
  * Virological failures and early discontinuations of therapy due to adverse events will be also registered.

SUMMARY:
* Unexpected results were published in 2016 showed increased aggressiveness and rates of HCC recurrence after curative treatment of HCC in HCV patients treated by DAAs achieving SVR. On the other hand, the retrospective analysis of ANRS study, did not observe an increased risk of HCC recurrence after DAAs treatment in patients who underwent curative HCC treatment.
* Assess the recurrence rate of HCC in HCV infected patients with prior history of treated HCC who achieved rCR with and without administration of DAAs and assess the effect of its timing.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common primary cancer of the liver, represents more than 90% of primary liver cancers, and is one of the leading cause of cancer-related death worldwide, therefore, it is a major global health problem.

In 2017, it is estimated that 40,710 people in the united states will be diagnosed with liver cancer and intrahepatic duct cancer; 29,200 males and 11,510 females and approximately 28,920 deaths. Incidence rates of HCC are 3 times higher in males than in females.

In Egypt, the estimated number of liver cancer is increasing as it was 29,975 in 2015 and will be 35,320 in 2020, 41,513 in 2025 and 85,471 in 2050. Liver cancer is the most frequent cancer in Egypt as it represents about 24% of all cancers in Egypt.

Cirrhosis is an important risk factor for HCC, and may be caused by chronic viral hepatitis, alcohol, inherited metabolic diseases such as hemochromatosis or alpha-1-antitrypsin deficiency, and non-alcoholic fatty liver disease. All causes of cirrhosis may be complicated by carcinogenesis, but the risk is higher in patients with hepatitis infection. Overall, one-third of cirrhotic patients will develop HCC during their lifetime.

Worldwide, approximately 54% of all cases of HCC are associated with hepatitis B virus (HBV) infection, while 31% are due to hepatitis c virus (HCV) infection, while only 15% are associated with other causes.

The prevalence of HCV infection in Egypt is the highest in the world, so its long-term consequences is a major endemic medical health problem in Egypt. The most common HCV RNA genotype in Egypt is genotype 4, representing more than 85% of all HCV cases in Egypt.

The direct acting antivirals (DAAs) are specific to the HCV particle and aim to inhibit viral RNA replication by attacking some of the various enzymes involved in the RNA replication process, thereby inhibiting viral replication, and causing viral eradication (Muir, 2014).

The primary goal of HCV therapy is to cure the infection, i.e. to achieve a sustained virological response (SVR) which defined as undetectable HCV RNA 12 weeks or 24 weeks after treatment completion. More than 95% of patients have SVR using DAAs except for genotype 3 virus in cirrhotic patients where SVR is still insufficient.

In the last decades before the era of DAAs, it was reported that SVR is associated with a reduction in all-cause mortality, liver mortality, and a reduction in the risk of HCC, this was by several meta-analyses which have studied this issue and suggested that SVR is associated with a reduction in the incidence of HCC in the long-term.

However, most of these studies are observational and retrospective and were based on SVR achieved with interferon (IFN) based therapy. Whether the high rates of SVR achieved with new IFN-free regimens reduce the risk of recurrence following resection or ablation of HCC is currently debated.

The success of DAAs against hepatitis C is a major breakthrough in Hepatology. Till now, there are very few data on the benefits of DAA-based antiviral therapy in patients who have already developed HCC, since this specific population have not been included in the pivotal trials.

Unexpected results were published in 2016 showed increased aggressiveness and rates of HCC recurrence after curative treatment of HCC in HCV patients treated by DAAs achieving SVR, one is a multicenter study conducted in Spain, of 58 patients and the other is a single center study, was done in Italy, of 59 patients, recurrences were 28% and 29%, respectively.

These studies were criticized due to the small number of patients, their retrospective character and lack of control arms, nevertheless their observation should be taken as a note of caution and need a larger assessment.

On the other hand, the retrospective analysis of the France REcherche Nord&sud Sida-vih Hépatites (ANRS) study in France, did not observe an increased risk of HCC recurrence after DAAs treatment, in patients who underwent curative HCC treatment including liver transplantation.

In addition, it was found in the preliminary results of a prospective observational study of HCV-infected patients with HCC given DAAs that there was no HCC recurrence following curative treatment over a median follow-up period of 12 months after DAA use.

Interestingly, it was reported that a decreased HCC incidence in decompensated cirrhotic patients with SVR achieved by DAAs compared to patients without SVR.

The mechanism which explains the high rate of tumor recurrence after DAAs treatment is that microenvironment and viral induced inflammation play an essential role in chronic liver injury and tumor initiation. However, the immune system has also an anti-tumor effect. Thus, there is a complex and fragile equilibrium between a pro tumor and anti-tumor function of the immune system.

Some studies have suggested that DAA treatment could modify natural killer function and expression of interferon response gene. Therefore, the hypothesis is a dysregulation of the anti-tumor response after the sudden decrease of HCV viral load induced by DAAs which promotes tumor recurrence. However, this phenomenon was unlikely to occur in patients who received IFN due to the slowly developing antiviral effect of this cytokine coupled with its immune modulatory and anti-proliferative properties.

However, this mechanism is purely theoretical and no strong preclinical studies support this hypothesis, but the high rate of HCC recurrence after DAA treatments in patients with prior HCC suggests that a close follow-up of these patients remains mandatory as well as a reassessment of these observations in a prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Age: more than or equal to 18 years old.
* Confirmed HCV viremia by PCR.
* CHILD Pugh "A".
* HCC diagnosed by criteria according to AASLD guidelines.
* HCC patients should have been treated prior to randomization by resection, or ablation and achieving rCR.

Exclusion Criteria:

* Patients below 18 old.
* Patients with advanced liver condition.
* Patients known HBV or HIV infection.
* Prior history of liver transplantation.
* HCC treatment but without rCR before randomization
* Pregnancy and lactation.
* Patients with other malignancies other than HCC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | Follow up will be done from baseline for up to 24 months for detection of sustained HCC treatment,tumoral progression or denovo occurrence
  To compare the Recurrence Rate of HCC in the two main randomized arms (administration of DAAs "arm 1" and control arm "arm 2")

SECONDARY OUTCOMES:
effect of timing of administration of DAAs after achieving rCR as regard recurrence rate | Follow up will be done from baseline for up to 24 months
  To assess the effect of timing of administration of DAAs after achieving rCR as regard recurrence rate in the 2 sub-groups of arm 1 (administration of DAAs after 3 months from rCR "group A" and administration after 6 months "group B")
Identifications of predictive factors of HCC recurrence | Follow up will be done from baseline for up to 24 months
  Identifications of predictive factors of HCC recurrence in chronic HCV patients treated with DAAs and achieved SVR.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conti F, Buonfiglioli F, Scuteri A, Crespi C, Bolondi L, Caraceni P, Foschi FG, Lenzi M, Mazzella G, Verucchi G, Andreone P, Brillanti S. Early occurrence and recurrence of hepatocellular carcinoma in HCV-related cirrhosis treated with direct-acting antivirals. J Hepatol. 2016 Oct;65(4):727-733. doi: 10.1016/j.jhep.2016.06.015. Epub 2016 Jun 24. PMID 27349488
- [Background] Elgharably A, Gomaa AI, Crossey MM, Norsworthy PJ, Waked I, Taylor-Robinson SD. Hepatitis C in Egypt - past, present, and future. Int J Gen Med. 2016 Dec 20;10:1-6. doi: 10.2147/IJGM.S119301. eCollection 2017. PMID 28053553
- [Background] European Association For The Study Of The Liver; European Organisation For Research And Treatment Of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. J Hepatol. 2012 Apr;56(4):908-43. doi: 10.1016/j.jhep.2011.12.001. No abstract available. PMID 22424438
- [Background] European Association for the Study of the Liver. EASL Recommendations on Treatment of Hepatitis C 2016. J Hepatol. 2017 Jan;66(1):153-194. doi: 10.1016/j.jhep.2016.09.001. Epub 2016 Sep 22. No abstract available. PMID 27667367
- [Background] ANRS collaborative study group on hepatocellular carcinoma (ANRS CO22 HEPATHER, CO12 CirVir and CO23 CUPILT cohorts). Electronic address: stanislas.pol@aphp.fr. Lack of evidence of an effect of direct-acting antivirals on the recurrence of hepatocellular carcinoma: Data from three ANRS cohorts. J Hepatol. 2016 Oct;65(4):734-740. doi: 10.1016/j.jhep.2016.05.045. Epub 2016 Jun 7. PMID 27288051
- [Background] Nault JC, Colombo M. Hepatocellular carcinoma and direct acting antiviral treatments: Controversy after the revolution. J Hepatol. 2016 Oct;65(4):663-665. doi: 10.1016/j.jhep.2016.07.004. Epub 2016 Jul 12. No abstract available. PMID 27417216
- [Background] Torres HA, Vauthey JN, Economides MP, Mahale P, Kaseb A. Hepatocellular carcinoma recurrence after treatment with direct-acting antivirals: First, do no harm by withdrawing treatment. J Hepatol. 2016 Oct;65(4):862-864. doi: 10.1016/j.jhep.2016.05.034. Epub 2016 May 30. No abstract available. PMID 27255582